CLINICAL TRIAL: NCT07009743
Title: A Prospective, Multicenter Study of O-RADS MRI System on Early Detection of Ovarian Cancer
Brief Title: O-RADS MRI System on Early Detection of Ovarian Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Responsible Party: Sponsor
Other Study IDs: O-RADS MRI
Record Dates: First submitted 2025-05-21; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer (OvCa); Ovarian Cancer Metastatic
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI contrast-enhancing agents — All patients underwent standard pelvic MRI examinations (1.5T or 3T) with the following sequences: T2-weighted imaging (T2WI), T1-weighted imaging (T1WI) with and without fat suppression; axial, sagittal, and coronal post-contrast T1WI following intravenous administration of gadolinium-based contrast agents (GBCA); functional sequences including dynamic contrast-enhanced MRI (DCE-MRI) and diffusion-weighted imaging MRI (DWI-MRI). Enhancement sequences may be omitted if no adnexal masses were identified on T2WI, T1WI, or DWI sequences.

SUMMARY:
This study is designed to prospectively enroll individuals with suspected or potential risk of ovarian cancer across multiple centers. The investigation will implement rational optimization of the recommended imaging sequences and interpretation protocols within the standard Ovarian-Adnexal Reporting and Data System (O-RADS) MRI framework. By integrating comprehensive clinical parameters and histopathological correlations, we aim to validate the diagnostic efficacy and reproducibility of the optimized protocol against the standard O-RADS MRI system. The ultimate objective is to establish a refined methodology for accurately diagnosing early-stage or low-burden ovarian malignancies, thereby improving prognostic outcomes of patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting either of the following criteria based on initial diagnostic pelvic ultrasound findings (pelvic mass or pelvic effusion) suspicious for ovarian malignancy or at elevated risk for ovarian cancer:

  1. Postmenopausal women or females ≥45 years with pelvic mass or effusion on ultrasound;
  2. Postmenopausal women or females ≥45 years with serum CA125 ≥35 U/mL;
  3. Females ≥35 years with a confirmed family history of ovarian or breast carcinoma;
  4. Females ≥35 years harboring pathogenic/likely pathogenic BRCA1/2 germline mutations;
  5. Females ≥35 years with BRCA1/2 mutations, non-suspicious adnexal lesions on ultrasound but planning prophylactic adnexectomy with availability of serial pathological sectioning.

     ② Ability to comply with the study protocol and adhere to scheduled follow-up assessments.

     ③ Provision of written informed consent.

     Exclusion Criteria:
     * ① Pregnant individuals

       * Patients with histopathologically confirmed ovarian cancer

         * Ovarian malignancy diagnosed by PET-CT at this institution

           ④ Patients undergoing neoadjuvant chemotherapy for confirmed ovarian cancer

           ⑤ Claustrophobia precluding tolerance of MRI examination

           ⑥ Contraindications to MRI: cardiac pacemakers, ferromagnetic implants, or high-risk metallic foreign bodies

           ⑦ History of gadolinium-based contrast agent (GBCA) hypersensitivity or intolerance

           ⑧ Severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73 m²)

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with epithelial ovarian carcinoma (EOC) at FIGO stages I-IIB and stage IIIC (with a tumor burden score <2).
Sampling Method: Probability Sample
Enrollment: 2549 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
the diagnostic performance of the O-RADS MRI system in the early detection of ovarian cancer | 2 years
  To evaluate the diagnostic performance of the O-RADS MRI system in the early detection of ovarian cancer (FIGO stages I-IIIC, epithelial ovarian carcinoma [EOC], tumor burden score ≤2), including sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), accuracy, and area under the receiver operating characteristic curve (AUC).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China, China